CLINICAL TRIAL: NCT00954447
Title: A Phase III Randomised, Double-blind, Placebo-controlled, Parallel Group Efficacy and Safety Study of Linagliptin (5 mg), Administered Orally Once Daily for at Least 52 Weeks in Type 2 Diabetic Patients in Combination With Basal Insulin Therapy
Brief Title: Efficacy and Safety of Linagliptin in Combination With Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.36; 2008-008296-33 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2012-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- Linagliptin (Experimental): patient receives a tablet with intended final marketed dose
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): patient receives a tablet identical to those containing Linagliptin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo, identical to Linagliptin tablet
  Arms: Placebo
Drug: Linagliptin — intended final marketed dose
  Arms: Linagliptin

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of linagliptin (5 mg / once daily) compared to Placebo during long term treatment (52 weeks and longer) in combination with basal insulin in patients with type 2 diabetes mellitus with insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

1. Diabetes type 2, detectable C-peptide, HbA1c 7-10%
2. Pretreatment with basal insulin +/- Metformin or/and +/- Pioglitazone 3 Age > 18 years, BMI <= 45 kg/m2

Exclusion criteria:

1. Uncontrolled hyperglycemia during Run-in
2. Myocardial infarction, stroke or TIA within 3 months prior to informed consent
3. Liver impairment; gastric surgery; medical history of cancer in last 5 years
4. Other antidiabetic drugs, antiobesity drugs, systemic steroids, other investigational drug before randomisation
5. Unsufficient birth control, pregnancy and nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1263 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (169):
- United States (47):
  - 1218.36.01043 Boehringer Ingelheim Investigational Site, Escondido, California
  - 1218.36.01051 Boehringer Ingelheim Investigational Site, Escondido, California
  - 1218.36.01065 Boehringer Ingelheim Investigational Site, Fresno, California
  - 1218.36.01021 Boehringer Ingelheim Investigational Site, Greenbrae, California
  - 1218.36.01013 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1218.36.01048 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1218.36.01058 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1218.36.01008 Boehringer Ingelheim Investigational Site, Santa Ana, California
  - 1218.36.01056 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1218.36.01054 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1218.36.01035 Boehringer Ingelheim Investigational Site, Inverness, Florida
  - 1218.36.01010 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.36.01042 Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - 1218.36.01063 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1218.36.01037 Boehringer Ingelheim Investigational Site, Ponte Vedra, Florida
  - 1218.36.01032 Boehringer Ingelheim Investigational Site, Saint Cloud, Florida
  - 1218.36.01049 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1218.36.01036 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1218.36.01047 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1218.36.01009 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 1218.36.01055 Boehringer Ingelheim Investigational Site, Honolulu, Hawaii
  - 1218.36.01014 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1218.36.01011 Boehringer Ingelheim Investigational Site, Paducah, Kentucky
  - 1218.36.01034 Boehringer Ingelheim Investigational Site, City of Saint Peters, Missouri
  - 1218.36.01040 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1218.36.01029 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1218.36.01018 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1218.36.01053 Boehringer Ingelheim Investigational Site, New Hartford, New York
  - 1218.36.01006 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1218.36.01025 Boehringer Ingelheim Investigational Site, Hickory, North Carolina
  - 1218.36.01005 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 1218.36.01015 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1218.36.01039 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1218.36.01019 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 1218.36.01012 Boehringer Ingelheim Investigational Site, Norristown, Pennsylvania
  - 1218.36.01004 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1218.36.01020 Boehringer Ingelheim Investigational Site, Simpsonville, South Carolina
  - 1218.36.01003 Boehringer Ingelheim Investigational Site, Kingsport, Tennessee
  - 1218.36.01038 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.36.01016 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.36.01026 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1218.36.01041 Boehringer Ingelheim Investigational Site, Bennington, Vermont
  - 1218.36.01064 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1218.36.01024 Boehringer Ingelheim Investigational Site, Lakewood, Washington
  - 1218.36.01007 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 1218.36.01027 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1218.36.01062 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Argentina (5):
  - 1218.36.54001 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.36.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.36.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.36.54005 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.36.54004 Boehringer Ingelheim Investigational Site, Córdoba
- Belgium (3):
  - 1218.36.32002 Boehringer Ingelheim Investigational Site, Edegem
  - 1218.36.320099 Boehringer Ingelheim Investigational Site, Edegem
  - 1218.36.32006 Boehringer Ingelheim Investigational Site, Sint-Gillis-Waas
- Brazil (4):
  - 1218.36.55003 Boehringer Ingelheim Investigational Site, Belém
  - 1218.36.55004 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1218.36.55001 Boehringer Ingelheim Investigational Site, São Paulo
  - 1218.36.55002 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (11):
  - 1218.36.02010 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.36.02004 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.36.02011 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1218.36.02006 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1218.36.02002 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1218.36.02009 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.36.02005 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 1218.36.02008 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.36.02007 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.36.02001 Boehringer Ingelheim Investigational Site, Laval, Quebec
  - 1218.36.02003 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Czechia (6):
  - 1218.36.42004 Boehringer Ingelheim Investigational Site, Brno
  - 1218.36.42006 Boehringer Ingelheim Investigational Site, Břeclav
  - 1218.36.42005 Boehringer Ingelheim Investigational Site, Hodonín
  - 1218.36.42002 Boehringer Ingelheim Investigational Site, Mladá Boleslav
  - 1218.36.42001 Boehringer Ingelheim Investigational Site, Neratovice
  - 1218.36.42007 Boehringer Ingelheim Investigational Site, Zlín
- Finland (6):
  - 1218.36.35807 Boehringer Ingelheim Investigational Site, Joensuu
  - 1218.36.35802 Boehringer Ingelheim Investigational Site, Kuopio
  - 1218.36.35803 Boehringer Ingelheim Investigational Site, Oulu
  - 1218.36.35805 Boehringer Ingelheim Investigational Site, Tampere
  - 1218.36.35804 Boehringer Ingelheim Investigational Site, Turku
  - 1218.36.35806 Boehringer Ingelheim Investigational Site, Vantaa
- Germany (16):
  - 1218.36.49001 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.36.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.36.49010 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.36.49009 Boehringer Ingelheim Investigational Site, Bosenheim
  - 1218.36.49017 Boehringer Ingelheim Investigational Site, Cologne
  - 1218.36.49004 Boehringer Ingelheim Investigational Site, Dortmund
  - 1218.36.49006 Boehringer Ingelheim Investigational Site, Dresden
  - 1218.36.49012 Boehringer Ingelheim Investigational Site, Magdeburg
  - 1218.36.49005 Boehringer Ingelheim Investigational Site, Mainz
  - 1218.36.49018 Boehringer Ingelheim Investigational Site, Neuwied
  - 1218.36.49008 Boehringer Ingelheim Investigational Site, Pirna
  - 1218.36.49019 Boehringer Ingelheim Investigational Site, Sulzbach-Rosenberg
  - 1218.36.49003 Boehringer Ingelheim Investigational Site, Unterschneidheim
  - 1218.36.49011 Boehringer Ingelheim Investigational Site, Wangen
  - 1218.36.49014 Boehringer Ingelheim Investigational Site, Wangen
  - 1218.36.49015 Boehringer Ingelheim Investigational Site, Westerkappeln
- Greece (6):
  - 1218.36.30003 Boehringer Ingelheim Investigational Site, Athens
  - 1218.36.30007 Boehringer Ingelheim Investigational Site, Athens
  - 1218.36.30010 Boehringer Ingelheim Investigational Site, Athens
  - 1218.36.30011 Boehringer Ingelheim Investigational Site, Larissa
  - 1218.36.30002 Boehringer Ingelheim Investigational Site, Nikaia
  - 1218.36.30005 Boehringer Ingelheim Investigational Site, Thessaloniki
- Italy (7):
  - 1218.36.39002 Boehringer Ingelheim Investigational Site, Ferrara
  - 1218.36.39003 Boehringer Ingelheim Investigational Site, Ferrara
  - 1218.36.39004 Boehringer Ingelheim Investigational Site, Genova
  - 1218.36.39005 Boehringer Ingelheim Investigational Site, Milan
  - 1218.36.39001 Boehringer Ingelheim Investigational Site, Pordenone
  - 1218.36.39007 Boehringer Ingelheim Investigational Site, Siena
  - 1218.36.39006 Boehringer Ingelheim Investigational Site, Syracuse
- Mexico (3):
  - 1218.36.52002 Boehringer Ingelheim Investigational Site, Pachuca
  - 1218.36.52004 Boehringer Ingelheim Investigational Site, San Luis Potosí City
  - 1218.36.52005 Boehringer Ingelheim Investigational Site, Tijuana
- Netherlands (7):
  - 1218.36.31008 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1218.36.31001 Boehringer Ingelheim Investigational Site, Almere Stad
  - 1218.36.31006 Boehringer Ingelheim Investigational Site, Beek
  - 1218.36.31002 Boehringer Ingelheim Investigational Site, Ewijk
  - 1218.36.31004 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1218.36.31007 Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - 1218.36.31005 Boehringer Ingelheim Investigational Site, Wildervank
- Norway (5):
  - 1218.36.47002 Boehringer Ingelheim Investigational Site, Bergen
  - 1218.36.47006 Boehringer Ingelheim Investigational Site, Elverum
  - 1218.36.47005 Boehringer Ingelheim Investigational Site, Hamar
  - 1218.36.47004 Boehringer Ingelheim Investigational Site, Oslo
  - 1218.36.47001 Boehringer Ingelheim Investigational Site, Stavanger
- 1218.36.51003 Boehringer Ingelheim Investigational Site, Lima, Peru
- Russia (6):
  - 1218.36.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.36.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.36.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.36.70001 Boehringer Ingelheim Investigational Site, Samara
  - 1218.36.70007 Boehringer Ingelheim Investigational Site, Smolensk
  - 1218.36.70006 Boehringer Ingelheim Investigational Site, Yaroslavl
- Slovakia (6):
  - 1218.36.42103 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1218.36.42101 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.36.42102 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.36.42104 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.36.42105 Boehringer Ingelheim Investigational Site, Prešov
  - 1218.36.42106 Boehringer Ingelheim Investigational Site, Trebišov
- South Korea (10):
  - 1218.36.82004 Boehringer Ingelheim Investigational Site, Daegu
  - 1218.36.82009 Boehringer Ingelheim Investigational Site, Daegu
  - 1218.36.82008 Boehringer Ingelheim Investigational Site, Incheon
  - 1218.36.82007 Boehringer Ingelheim Investigational Site, Jeonju
  - 1218.36.82001 Boehringer Ingelheim Investigational Site, Pusan
  - 1218.36.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.36.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.36.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.36.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.36.82010 Boehringer Ingelheim Investigational Site, Suwon
- Spain (10):
  - 1218.36.34002 Boehringer Ingelheim Investigational Site, Badia Del Vallés (Barcelona)
  - 1218.36.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 1218.36.34010 Boehringer Ingelheim Investigational Site, Barcelona
  - 1218.36.34001 Boehringer Ingelheim Investigational Site, Bercelona
  - 1218.36.34007 Boehringer Ingelheim Investigational Site, Borges Del Camp (Tarragona)
  - 1218.36.34003 Boehringer Ingelheim Investigational Site, Centelles (Barcelona)
  - 1218.36.34004 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1218.36.34011 Boehringer Ingelheim Investigational Site, Seville
  - 1218.36.34009 Boehringer Ingelheim Investigational Site, Tàrrega (Lleida)
  - 1218.36.34006 Boehringer Ingelheim Investigational Site, Vic (Barcelona)
- Taiwan (10):
  - 1218.36.88610 Boehringer Ingelheim Investigational Site, Changhua
  - 1218.36.88607 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1218.36.88601 Boehringer Ingelheim Investigational Site, Taichung
  - 1218.36.88603 Boehringer Ingelheim Investigational Site, Taichung
  - 1218.36.88606 Boehringer Ingelheim Investigational Site, Tainan
  - 1218.36.88602 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.36.88604 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.36.88605 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.36.88608 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.36.88609 Boehringer Ingelheim Investigational Site, Taipei

REFERENCES:
- [Derived] Sheu WH, Park SW, Gong Y, Pinnetti S, Bhattacharya S, Patel S, Seck T, Woerle HJ. Linagliptin improves glycemic control after 1 year as add-on therapy to basal insulin in Asian patients with type 2 diabetes mellitus. Curr Med Res Opin. 2015 Mar;31(3):503-12. doi: 10.1185/03007995.2015.1010638. Epub 2015 Feb 13. PMID 25629790
- [Derived] Yki-Jarvinen H, Rosenstock J, Duran-Garcia S, Pinnetti S, Bhattacharya S, Thiemann S, Patel S, Woerle HJ. Effects of adding linagliptin to basal insulin regimen for inadequately controlled type 2 diabetes: a >/=52-week randomized, double-blind study. Diabetes Care. 2013 Dec;36(12):3875-81. doi: 10.2337/dc12-2718. Epub 2013 Sep 23. PMID 24062327

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomised, double-blind, placebo-controlled, parallel group study. Whilst 1263 were randomised, only 1261 were treated.
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo, orally taken, once daily. During the first 24 weeks of the randomised treatment period, the background dose of basal insulin and/or oral antidiabetic agents was to remain stable. From 24 weeks after randomisation until the end of the trial, adjustments to the dose of basal insulin (but not oral antidiabetic agents) were permitted.
- Linagliptin 5 mg: Patients randomized to receive treatment with Linagliptin 5mg, orally taken, once daily. During the first 24 weeks of the randomised treatment period, the background dose of basal insulin and/or oral antidiabetic agents was to remain stable. From 24 weeks after randomisation until the end of the trial, adjustments to the dose of basal insulin (but not oral antidiabetic agents) were permitted.
Period: Overall Study
Arm/Group | Placebo | Linagliptin 5 mg
Started | 630 | 631
Completed | 520 | 543
Not Completed | 110 | 88
Not completed — Adverse Event | 33 | 25
Not completed — Lack of Efficacy | 17 | 3
Not completed — Protocol Violation | 5 | 7
Not completed — Lost to Follow-up | 8 | 14
Not completed — Withdrawal by Subject | 26 | 21
Not completed — Other | 21 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 5 mg | Total
Number analyzed (Participants) | 630 | 631 | 1261
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (10.0) | 59.7 (9.9) | 60.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301 | 302 | 603
  Male | 329 | 329 | 658
Baseline HbA1c [Mean (Standard Deviation); unit: Percentage] — Baseline HbA1c was defined as the last available HbA1c measurement prior to the start of randomised study treatment.There were 617 patients with non-missing baseline HbA1c in Placebo group and 618 patients with non-missing values in Linagliptin 5 mg.
  Percentage | 8.29 (0.85) | 8.31 (0.85) | 8.30 (0.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c After 24 Weeks
Description: HbA1c is measured as a percentage. Adjusted for treatment, baseline HbA1c, categorical renal function impairment and concomitant Oral antidiabetic drugs (OAD)
Time Frame: Baseline and 24 weeks
Population: The Full Analysis Set (FAS) with a last observation carried forward (LOCF) approach. The FAS comprises all randomised patients who were treated with at least one dose of study medication, had a baseline HbA1c measurement, and had at least one on-treatment HbA1c measurement within the first 24 weeks of double-blind treatment.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Percentage | 0.07 (0.08) | -0.58 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.65, 95% CI [-0.74 to -0.55], Standard Error of Mean 0.05 — Linagliptin 5mg - Placebo

2. Secondary Outcome: Number of Patients With HbA1c < 7.0 Percent
Time Frame: 24 and 52 weeks
Population: FAS using the non-completers considered failure (NCF) approach, in which missing data due to premature discontinuation of a patient were considered as failure.
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Participants
  after 24 weeks of treatment | 56 | 134
  after 52 weeks of treatment | 44 | 109
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; FAS with baseline HbA1c >= 7.0 percent (NCF); there are 593 available values for Placebo and 595 for Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression of HbA1c < 7.0 percent at week 52; Odds Ratio (OR) = 2.935, 95% CI [1.949 to 4.419] — Linagliptin 5mg vs. Placebo OR adjusted for baseline HbA1c, categorical renal function impairment, concomitant OADs and treatment

3. Secondary Outcome: Number of Patients Lowering HbA1c by at Least 0.5 Percent
Time Frame: 24 and 52 weeks
Population: FAS (NCF)
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Participants
  after 24 weeks of treatment | 137 | 333
  after 52 weeks of treatment | 104 | 231

4. Secondary Outcome: Change From Baseline in HbA1c by Visit at Week 6
Description: Means adjusted for treatment, baseline HbA1c, categorical renal function impairment and concomitant OADs
Time Frame: Baseline and 6 weeks
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Percentage | 0.00 (0.05) | -0.45 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI [-0.51 to -0.39], Standard Error of Mean 0.03 — Linagliptin 5mg - Placebo

5. Secondary Outcome: Change From Baseline in HbA1c by Visit at Week 12
Description: Means adjusted for treatment, baseline HbA1c, categorical renal function impairment and concomitant OADs
Time Frame: Baseline and 12 weeks
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Percentage | 0.02 (0.07) | -0.59 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.61, 95% CI [-0.69 to -0.52], Standard Error of Mean 0.04 — Linagliptin 5mg - Placebo

6. Secondary Outcome: Change From Baseline in HbA1c by Visit at Week 18
Description: Means adjusted for treatment, baseline HbA1c, categorical renal function impairment and concomitant OADs
Time Frame: Baseline and 18 weeks
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Percentage | 0.03 (0.08) | -0.64 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.67, 95% CI [-0.76 to -0.57], Standard Error of Mean 0.05 — Linagliptin 5mg - Placebo

7. Secondary Outcome: Change From Baseline in HbA1c by Visit at Week 32
Description: Means adjusted for treatment, baseline HbA1c, categorical renal function impairment and concomitant OADs
Time Frame: Baseline and 32 weeks
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Percentage | 0.01 (0.08) | -0.56 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI [-0.67 to -0.47], Standard Error of Mean 0.05 — Linagliptin 5mg - Placebo

8. Secondary Outcome: Change From Baseline in HbA1c by Visit at Week 40
Description: Means adjusted for treatment, baseline HbA1c, categorical renal function impairment and concomitant OADs
Time Frame: Baseline and 40 weeks
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Percentage | 0.05 (0.08) | -0.50 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI [-0.65 to -0.45], Standard Error of Mean 0.05 — Linagliptin 5mg - Placebo

9. Secondary Outcome: Change From Baseline in HbA1c by Visit at Week 52
Description: Means adjusted for treatment, baseline HbA1c, categorical renal function impairment and concomitant OADs
Time Frame: Baseline and 52 weeks
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Percentage | 0.05 (0.08) | -0.48 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.53, 95% CI [-0.64 to -0.43], Standard Error of Mean 0.05 — Linagliptin 5mg - Placebo

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at 24 Weeks of Treatment
Description: Means adjusted for treatment, baseline HbA1c, baseline FPG, categorical renal function impairment and concomitant OADs
Time Frame: Baseline and 24 weeks
Population: FAS (LOCF), further restricted to patients with a baseline FPG measurement and at least one on-treatment FPG measurement
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 609 | 614
mg/dL | 4.52 (3.94) | -7.09 (3.97)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -11.60, 95% CI [-16.49 to -6.71], Standard Error of Mean 2.49 — Linagliptin 5mg - Placebo

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 52 Weeks of Treatment
Time Frame: Baseline and 52 weeks
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 609 | 614
mg/dL | 0.63 (56.44) | -2.55 (55.01)

12. Secondary Outcome: Change From Baseline in FPG
Time Frame: Baseline, 6, 12, 18, 24, 32 and 40 weeks
Population: FAS, observed cases (OC)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 600 | 606
mg/dL
  after 6 weeks of treatment | 2.97 (50.89) | -5.29 (44.74)
  after 12 weeks of treatment (N=556, N=590) | -0.33 (51.09) | -7.59 (48.50)
  after 18 weeks of treatment (N=533, N=567) | 2.10 (53.21) | -3.30 (55.51)
  after 24 weeks of treatment (N=499, N=533) | 0.04 (54.94) | -7.07 (44.70)
  after 32 weeks of treatment (N=436, N=491) | -2.67 (52.43) | -6.30 (48.16)
  after 40 weeks of treatment (N=357, N=429) | -3.99 (50.29) | -6.50 (50.00)

13. Secondary Outcome: Change From Baseline in Mean Insulin Dose at 52 Weeks of Treatment
Description: Means adjusted for treatment, continous baseline HbA1c, continous baseline weight, continous baseline Insulin, categorical renal function impairment and concomitant OADs
Time Frame: Baseline and 52 weeks
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: International units (IU)
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
International units (IU) | 4.18 (0.84) | 2.60 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p = 0.0029, ANCOVA; Mean Difference (Final Values) = -1.58, 95% CI [-2.61 to -0.54], Standard Error of Mean 0.53 — Linagliptin 5mg - Placebo

14. Secondary Outcome: Change From Baseline in Weighted Mean Daily Glucose After 24 and 52 Weeks of Treatment
Description: Mean Daily Glucose was calculated using the 8-point blood glucose profile
Time Frame: Baseline, 24 and 52 weeks
Population: FAS (OC)
Measure: Mean (Standard Deviation); unit: mmol*hr/L
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 55 | 52
mmol*hr/L
  after 24 weeks of treatment | 0.03 (2.28) | -0.01 (1.98)
  after 52 weeks of treatment (N=25, N=15) | 0.10 (3.06) | -0.50 (2.35)

15. Secondary Outcome: Change From Baseline in Incremental Post-prandial Glucose (iPPG) After 24 Weeks of Treatment
Time Frame: Baseline and 24 weeks: post-breakfast, post-lunch, post-dinner
Population: FAS (OC)
Measure: Mean (Standard Deviation); unit: mmol*hr/L
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 60 | 61
mmol*hr/L
  post-breakfast incremental glucose | 9.31 (44.02) | -3.78 (63.63)
  post-lunch incremental glucose (N=34, N=41) | -17.80 (61.94) | -11.00 (68.04)
  post-dinner incremental glucose (N=46, N=57) | -1.71 (68.15) | -3.26 (66.51)

16. Other Pre Specified Outcome: Number of Patients With HbA1c < 6.5 Percent
Time Frame: 24 and 52 weeks
Population: FAS (NCF)
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 617 | 618
Participants
  after 24 weeks of treatment | 10 | 50
  after 52 weeks of treatment | 12 | 46
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; FAS with baseline HbA1c >= 6.5 percent (NCF); there are 615 available values for Placebo and 616 for Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Logistic regression of HbA1c < 6.5 percent at week 52; Odds Ratio (OR) = 4.327, 95% CI [2.221 to 8.430] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Placebo | Linagliptin 5 mg
Serious Adverse Events (participants affected / at risk) | 83/630 | 87/631
Other Adverse Events (participants affected / at risk) | 354/630 | 354/631
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=630) | Linagliptin 5 mg (N=631)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 2
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Diplopia (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 0
Retinopathy proliferative (Eye disorders) | 1 | 0
Vitreous adhesions (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 2
Infected skin ulcer (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Meningitis streptococcal (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Electric shock (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Colonoscopy (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Ureteral catheterisation (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=630) | Linagliptin 5 mg (N=631)
Diarrhoea (Gastrointestinal disorders) | 30 | 33
Influenza (Infections and infestations) | 33 | 26
Nasopharyngitis (Infections and infestations) | 62 | 71
Urinary tract infection (Infections and infestations) | 43 | 30
Hyperglycaemia (Metabolism and nutrition disorders) | 112 | 90
Hypoglycaemia (Metabolism and nutrition disorders) | 197 | 191
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 34
Dizziness (Nervous system disorders) | 30 | 33
Headache (Nervous system disorders) | 27 | 35
Hypertension (Vascular disorders) | 35 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.